CLINICAL TRIAL: NCT03212690
Title: Study to Elucidate the Association of the Renin-angiotensin System and Right Ventricular Function in Mechanically Ventilated Patients
Brief Title: Study of Renin-angiotensin System in Mechanically Ventilated Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study stopped early following termination of associated clinical development program (due to lack of efficacy)
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 205821; 2017-A01653-50 (Registry Identifier: Biological Research and Collections)
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Results first posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Acute Lung Injury
Keywords: mechanical ventilation; echocardiography; right ventricular function; Ang (1-7); Ang II; Renin-angiotensin system
MeSH Terms: conditions — Acute Lung Injury | interventions — Respiration, Artificial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mechanically ventilated subjects (Experimental): Subjects receiving invasive mechanical ventilation (Duration of ventilation <=48 hours) will be evaluated using standard care investigations.
  Interventions: Drug: Local standard of care; Procedure: Mechanical ventilation

INTERVENTIONS:
Drug: Local standard of care — Local standard of care will include fluid resuscitation, use of vasopressor drugs and renal support.
Procedure: Mechanical ventilation — Mechanical ventilation will be based on volume-assist control mode, with a target tidal volume of 6-8 milliliter per kg (mL/kg) and a target plateau pressure of 30 centimeter of water (cmH2O).

SUMMARY:
The purpose of this study is to assess whether circulating Angiotensin (Ang) II and Ang (1-7) levels are associated with right ventricular (RV) dysfunction in mechanically ventilated subjects. It is also designed to further characterize the subject population for severity of RV dysfunction. This study will investigate the association of renin-angiotensin system (RAS) peptides and markers of RV function, as measured by echocardiography, in subjects requiring acute mechanical ventilation. Maximum 150 subjects will be enrolled for the study and they will be evaluated over three days period using standard of care investigations, including trans-thoracic echocardiography (TTE) and/or trans-esophageal echocardiography (TOE) echocardiography. The maximum total duration of this study for subjects is 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject must be 18 to 80 years of age inclusive, at the time of enrolment.
* Subjects who are receiving invasive mechanical ventilation (duration of ventilation less than equal to 48 hours).
* Body mass index within the range 18.0 - 38.0 kilograms per meter square (kg/m^2, inclusive). Clinical estimate of height and weight is acceptable.
* Given subjects will be mechanically ventilated upon enrolment, obtaining informed consent directly from the subjects will not be feasible. Consent will be obtained by subject's Legally Acceptable Representative (LAR) or subject will be enrolled upon emergency consent process or subject will be enrolled by signing the informed consent.

Exclusion Criteria:

* Subjects who are moribund or whose clinical condition is deteriorating rapidly or any subject for whom the investigator does not consider there is a reasonable expectation that they will be able to complete the 3 days of observation in the study.
* Subjects undergoing elective surgery. Investigator will make every effort to ensure that the following exclusion criteria are met; however, in some instances it may not be possible to assess all of these criteria within the 48-hour window. In this case, a subject can be included and investigator will obtain the information when available.
* Chronic obstructive pulmonary disease (COPD) requiring long term oxygen treatment or home mechanical ventilation.
* Documented pre-existing chronic pulmonary hypertension.
* Massive pulmonary embolism (defined by pulmonary embolism with systemic hypotension [defined as a systolic arterial pressure less than 90 mmHg or a drop in systolic arterial pressure of at least 40 mmHg for at least 15 minutes (mins)] which is not caused by new onset arrhythmias) or shock (manifested by evidence of tissue hypo-perfusion and hypoxia, including an altered level of consciousness, oliguria, or cool, clammy extremities).
* Pulmonary vasculitis or pulmonary hemorrhage including diffuse alveolar hemorrhage.
* Lung transplantation within last 6 months.
* Cardiopulmonary arrest during concurrent illness.
* Any use of RAS modulators including Angiotensin Converting Enzyme (ACE) type 1 inhibitors, Renin inhibitors and Angiotensin Receptor Blockers within 4 days or 5.5 half live whichever is longer.
* Do not resuscitate status.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- France (2):
  - GSK Investigational Site, Boulogne-Billancourt
  - GSK Investigational Site, Créteil

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted when justified, for up to another 12 months
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study elucidated the association of the Renin-angiotensin system and right ventricular (RV) function in mechanically ventilated participants. This study was conducted at two centers in France from 11-June-2018 to 08-July-2019. A total of 57 participants were enrolled in this study.
Pre-assignment Details: The study was terminated as overall probability of project success was considered low. The study had significant programmatic risks identified with development plan for Recombinant Human Angiotensin Converting Enzyme2 in critical care including participant identification, uncertainty around potential to impact mortality and operational feasibility.
Groups:
- Mechanically Ventilated Participants: Participants were enrolled following being mechanically ventilated and had their first echocardiogram (transthoracic echocardiogram [TTE] and transoesophageal echocardiogram [TOE]) within 48 hours of mechanical ventilation. Participants were assessed every 24 hours for a further two days with daily echocardiography to monitor right and left ventricular function. Participants received standard of care including fluid, use of vasopressor drugs and renal support.
Period: Overall Study
Arm/Group | Mechanically Ventilated Participants
Started | 57
Completed | 56
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Mechanically Ventilated Participants: Participants were enrolled following being mechanically ventilated and had their first echocardiogram (TTE and TOE) within 48 hours of mechanical ventilation. Participants were assessed every 24 hours for a further two days with daily echocardiography to monitor right and left ventricular function. Participants received standard of care including fluid, use of vasopressor drugs and renal support.
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.74 (12.807)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 57

OUTCOME MEASURES:

1. Primary Outcome: Renin-angiotensin System Cascade Biomarker to Include Angiotensin (Ang) II Level
Description: Blood samples were collected for renin-angiotensin system biomarkers at indicated time points. Evaluable Population consisted of all participants for whom pulmonary arterial systolic pressure (PASP), ratio of right ventricular to left ventricular end-diastolic area (RV size ratio), Ang II and Ang(1-7) data have been recorded for at least one study time point, and who did not retrospectively withdraw the consent.
Time Frame: Days 1, 2 and 3
Population: Evaluable Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 44
Picograms per milliliter
  Day 1, n=44 | 41.693 (67.4893)
  Day 2, n=43: number analyzed (Participants) | 43
  Day 2, n=43 | 43.861 (110.6191)
  Day 3, n=35: number analyzed (Participants) | 35
  Day 3, n=35 | 27.801 (49.1054)

2. Primary Outcome: Ratio of RV to Left Ventricular (LV) End-diastolic Area (RV Size Ratio)
Description: Right ventricular size ratio was measured using TTE or TOE.
Time Frame: Days 1, 2 and 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 45
Ratio
  Day 1, n=45 | 0.653 (0.2418)
  Day 2, n=42: number analyzed (Participants) | 42
  Day 2, n=42 | 0.655 (0.2276)
  Day 3, n=35: number analyzed (Participants) | 35
  Day 3, n=35 | 0.634 (0.1662)

3. Primary Outcome: Number of Participants With Paradoxical Septal Motion
Description: Paradoxical septal motion is the systolic movement of the interventricular septum toward the RV despite normal thickening. Paradoxical septal motion was measured by TTE or TOE. Number of participants who had paradoxical septal motion have been reported.
Time Frame: Days 1, 2 and 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 43
Participants
  Day 1, n=43 | 5
  Day 2, n=41: number analyzed (Participants) | 41
  Day 2, n=41 | 11
  Day 3, n=34: number analyzed (Participants) | 34
  Day 3, n=34 | 10

4. Primary Outcome: Pulmonary Arterial Systolic Pressure at Indicated Time Points
Description: Pulmonary arterial systolic pressure was measured using TTE or TOE.
Time Frame: Days 1, 2 and 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 39
Millimeters of mercury
  Day 1, n=38: number analyzed (Participants) | 38
  Day 1, n=38 | 36.350 (15.7070)
  Day 2, n=39 | 35.564 (12.2985)
  Day 3, n=29: number analyzed (Participants) | 29
  Day 3, n=29 | 37.224 (13.3521)

5. Primary Outcome: Right Atrial Pressure at Indicated Time Points
Description: Right atrial pressure is the blood pressure in the right atrium of the heart. Right atrial pressure was measured by TTE or TOE.
Time Frame: Days 1, 2 and 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 42
Millimeters of mercury
  Day 1, n=42 | 9.055 (4.5279)
  Day 2, n=40: number analyzed (Participants) | 40
  Day 2, n=40 | 9.425 (5.0530)
  Day 3, n=34: number analyzed (Participants) | 34
  Day 3, n=34 | 9.456 (4.7456)

6. Primary Outcome: Inferior Vena Cava Diameter at End Expiration at Indicated Time Points
Description: Inferior vena cava diameter was measured using TTE or TOE. Pulmonary arterial systolic pressure was estimated from trans-tricuspid pressure and right atrial pressure or inferior vena cava diameter.
Time Frame: Days 1, 2 and 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeter
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 41
Millimeter
  Day 1, n=38: number analyzed (Participants) | 38
  Day 1, n=38 | 18.529 (4.8940)
  Day 2, n=41 | 18.412 (5.5483)
  Day 3, n=34: number analyzed (Participants) | 34
  Day 3, n=34 | 17.915 (5.0126)

7. Primary Outcome: Pearson Correlation Coefficient Between PASP and Ang II Level
Description: Pearson correlation coefficient between PASP and Ang II level was derived using all available data from participants in the evaluable population. Pearson's correlation coefficient is a measure of the linear dependence between 2 variables. A correlation of +1 or -1 may occur if the data from the 2 variables lie exactly on a line. Pearson's correlation coefficient was calculated using Statistical Analysis Software (SAS).
Time Frame: Up to Day 3
Population: Evaluable Population.
Measure: Number; unit: Unitless
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 45
Unitless | -0.019

8. Primary Outcome: Pearson Correlation Coefficient Between RV Size Ratio and Ang II Level
Description: Pearson correlation coefficient between RV size ratio and Ang II level was derived using all available data from participants in the evaluable population. Pearson's correlation coefficient is a measure of the linear dependence between 2 variables. A correlation of +1 or -1 may occur if the data from the 2 variables lie exactly on a line. Pearson's correlation coefficient was calculated using SAS.
Time Frame: Up to Day 3
Population: Evaluable Population.
Measure: Number; unit: Unitless
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 45
Unitless | 0.153

9. Secondary Outcome: Number of Participants With Pulmonary Circulatory Dysfunction
Description: Pulmonary circulatory dysfunction is defined as moderate dysfunction (pulmonary arterial systolic pressure [>40 millimeters of mercury] or a dilated RV end diastolic RV/left ventricle [LV] area ratio [>=0.6] but without septal dyskinesia). At risk Population consisted of participants who satisfied following criteria: 1. pulmonary arterial systolic pressure and ratio of RV to LV end-diastolic area recorded for all three study days [regardless of the Ang II and Ang(1-7) status] and/or; 2. databased acute cor pulmonale/pulmonary circulatory dysfunction and/or acute respiratory distress syndrome (ARDS) assessment during the study period (even if they do not have three days worth of study assessments for the echo outcomes) were evaluated for acute cor pulmonale/pulmonary circulatory dysfunction and ARDS incidence rates. Number of participants with Pulmonary Circulatory Dysfunction have been reported.
Time Frame: Days 1, 2 and 3
Population: At risk Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 56
Participants
  Day 1, n=56 | 18
  Day 2, n=52: number analyzed (Participants) | 52
  Day 2, n=52 | 12
  Day 3, n=43: number analyzed (Participants) | 43
  Day 3, n=43 | 5

10. Secondary Outcome: Number of Participants With Acute Cor Pulmonale
Description: Acute cor pulmonale is defined as a dilated RV in the mid-esophagus longitudinal view or apical 4-chamber view (end-diastolic RV/LV area ratio [0.6]) associated with the presence of a septal dyskinesia in the (transgastric) short-axis view of the heart. Number of participants with acute cor pulmonale have been reported.
Time Frame: Days 1, 2 and 3
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 56
Participants
  Day 1, n=56 | 5
  Day 2, n=52: number analyzed (Participants) | 52
  Day 2, n=52 | 10
  Day 3, n=43: number analyzed (Participants) | 43
  Day 3, n=43 | 8

11. Secondary Outcome: Number of Participants With Severe Acute Cor Pulmonale
Description: Severe acute cor pulmonale is defined as severely dilated RV (end-diastolic RV/LV area ratio >=1) with septal dyskinesia. Number of participants with severe acute cor pulmonale have been reported.
Time Frame: Days 1, 2 and 3
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 56
Participants
  Day 1, n=56 | 3
  Day 2, n=52: number analyzed (Participants) | 52
  Day 2, n=52 | 0
  Day 3, n=43: number analyzed (Participants) | 43
  Day 3, n=43 | 0

12. Secondary Outcome: Renin-angiotensin System Cascade Biomarker: Ang(1-7) Level
Description: Blood samples were collected for renin-angiotensin system biomarkers at indicated time points.
Time Frame: Days 1, 2 and 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 44
Picograms per milliliter
  Day 1, n=44 | 6.038 (11.7629)
  Day 2, n=44 | 6.020 (11.3192)
  Day 3, n=36: number analyzed (Participants) | 36
  Day 3, n=36 | 4.911 (7.8364)

13. Secondary Outcome: Renin-angiotensin System Cascade Biomarker: Ang II/ Ang(1-7) Ratio
Description: Blood samples were collected for renin-angiotensin system biomarkers at indicated time points.
Time Frame: Days 1, 2 and 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 44
Ratio
  Day 1, n=44 | 10.620 (10.1424)
  Day 2, n=43: number analyzed (Participants) | 43
  Day 2, n=43 | 9.184 (7.3338)
  Day 3, n=35: number analyzed (Participants) | 35
  Day 3, n=35 | 7.938 (8.0332)

14. Secondary Outcome: Pearson Correlation Coefficient Between PASP and Ang(1-7)
Description: Pearson correlation coefficient between PASP and Ang(1-7) was derived using all available data from participants in the evaluable population. Pearson's correlation coefficient is a measure of the linear dependence between 2 variables. A correlation of +1 or -1 may occur if the data from the 2 variables lie exactly on a line. Pearson's correlation coefficient was calculated using SAS.
Time Frame: Up to Day 3
Population: Evaluable Population.
Measure: Number; unit: Unitless
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 45
Unitless | -0.050

15. Secondary Outcome: Pearson Correlation Coefficient Between PASP and Ang II/Ang(1-7)
Description: Pearson correlation coefficient between PASP and Ang II/Ang(1-7) was derived using all available data from participants in the evaluable population. Pearson's correlation coefficient is a measure of the linear dependence between 2 variables. A correlation of +1 or -1 may occur if the data from the 2 variables lie exactly on a line. Pearson's correlation coefficient was calculated using SAS.
Time Frame: Up to Day 3
Population: Evaluable Population.
Measure: Number; unit: Unitless
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 45
Unitless | 0.193

16. Secondary Outcome: Pearson Correlation Coefficient Between RV Size Ratio and Ang(1-7)
Description: Pearson correlation coefficient between RV size ratio and Ang(1-7) was derived using all available data from participants in the evaluable population. Pearson's correlation coefficient is a measure of the linear dependence between 2 variables. A correlation of +1 or -1 may occur if the data from the 2 variables lie exactly on a line. Pearson's correlation coefficient was calculated using SAS.
Time Frame: Up to Day 3
Population: Evaluable Population.
Measure: Number; unit: Unitless
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 45
Unitless | 0.350

17. Secondary Outcome: Pearson Correlation Coefficient Between RV Size Ratio and Ang II/Ang(1-7)
Description: Pearson correlation coefficient between RV size ratio and Ang II/Ang(1-7) was derived using all available data from participants in the evaluable population. Pearson's correlation coefficient is a measure of the linear dependence between 2 variables. A correlation of +1 or -1 may occur if the data from the 2 variables lie exactly on a line. Pearson's correlation coefficient was calculated using SAS.
Time Frame: Up to Day 3
Population: Evaluable Population.
Measure: Number; unit: Unitless
Arm/Group | Mechanically Ventilated Participants
Number analyzed (Participants) | 45
Unitless | -0.032

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events were collected up to Day 3
Description: Safety Population consisted of all participants for whom at least one echocardiograph and/or blood sample has been taken, and who did not retrospectively withdraw the consent.
Arm/Group | Mechanically Ventilated Participants
All-Cause Mortality (participants affected / at risk) | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57
Other Adverse Events (participants affected / at risk) | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-07-30): https://cdn.clinicaltrials.gov/large-docs/90/NCT03212690/SAP_000.pdf
  • Study Protocol (2019-02-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT03212690/Prot_001.pdf